CLINICAL TRIAL: NCT02852122
Title: The Role of C-11 Choline PET in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Chen Yen, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 102-3271A
Record Dates: First submitted 2015-07-08; First posted 2016-08-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Latent Cancer Prostate
Keywords: prostate cancer; C11 Choline PET/MR; staging; biochemical failure
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-11 choline (Experimental)
  Interventions: Drug: C-11 choline

INTERVENTIONS:
Drug: C-11 choline — This is an uncontrolled, open-labeled, non-randomized, prospective study. The study duration is expected to be completed in a period of 2 years. Up to 54 patients with primary prostate cancer and stratified as high risk group (PSA > 20 ng/mL, or Gleason score 8-10, or clinical stage >T2c) would be included.

SUMMARY:
The investigators determine the target number as 54 patients based on the following reasons: (a) The bony metastasis rate for the high risk prostate cancer patients with PSA from 20 to 99.9 ng/ml was 21% (166/767 cases in a systemic review) [8]; the estimated sample size would be 47 under the condition of 20% more distant metastasis cases were identified by the PET/MRI scan using the 90% power, significance level of 0.05 and one sample proportion test. Assuming a dropout rate of 10%, the final ideal sample size is 52 patients. (b) The newly diagnostic number for the high risk prostate cancer patients in our hospital annually is ~70, about 6 patients a month. It is clinically feasible to recruit 3 patients a month until 18 months since the study begin. The study could be completed in 2 years with 54 cases

DETAILED DESCRIPTION:
[11C] choline positron emission tomography (PET) is an emerging modality for staging at initial diagnosis or re-staging at the time of treatment failure. The updated study shows 11C -labeled choline derivatives seem to be the most promising PET radionuclides in assessment of prostate cancer and USA FDA approves the utility of C-11 Choline in prostate cancer patients in 2012 September.

To our best literature search, there are only few preliminary studies regarding application of PET/MR in prostate cancer patients and the initial results in correlation of functional MRI and PET images seems promising. Combined PET/MRI images have the advantage of giving anatomical, functional, and metabolic information in a single image setting and provide a comprehensive survey including local regional extension and systemic metastasis. Unlike in the USA where more than 70% prostate cancer patients were diagnosed at early stage, most prostate cancer patients in Taiwan were diagnosed at advanced stage with high PSA or T3-4 disease, or even systemic metastasis. The need to implement good staging modality is even more urgently needed in Taiwan than in USA and related studies are still lacking. In the current study, our hypothesis is that C-11 Choline PET/MRI is a good modality in staging high risk prostate cancer patients, and in predicting patients' outcome after treatment. Our hypothesis will be examined by this clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically suspicious and/or pathology-proved high risk group prostate cancer patients (PSA > 20 ng/mL, or Gleason score 8-10, or clinical stage >T2c)
2. Age equals or more than 20 years old
3. Willing to sign the informed consent

Exclusion Criteria:

1. Patients with a concomitant or previous malignancy history
2. Unable to tolerate MR or PET/CT scan, such as those with magnetic implants (e.g. those received intracranial aneurysm surgery, cardiac pacemaker, artificial valves replacement, artificial ears, hip prosthesis), claustrophobia, unable to lie still
3. Unable to give informed consent
4. Previous allergy to carbon-labelled radionuclide

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Role of C-11 Choline PET in Patients with Prostate Cancer | Two years
  Inconsistence rate (%) of C-11 Choline PET and MRI in detecting local regional and distant metastasis prostate cancer. The inconsistence rate (%) is defined as the proportion of inconsistent results by PET and MRI, i. e. PET positive but MRI negative, or PET negative but MRI positive.